CLINICAL TRIAL: NCT02002819
Title: Phase 2a Levetiracetam Trial for AD-Associated Network Hyperexcitability
Brief Title: Levetiracetam for Alzheimer's Disease-Associated Network Hyperexcitability
Acronym: LEV-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NEUR-2017-25879; PCTRB-13-288476 (Other Grant/Funding Number: Alzheimer's Association Inc.)
Record Dates: First submitted 2013-10-25; First posted 2013-12-06 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; AD; Early-onset AD; EOAD; Early-onset Alzheimer's; Early-onset Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam-Placebo (Experimental): This group receives levetiracetam for 4 weeks twice daily, then has a break where no treatment is given for 4 weeks, and then receives placebo for 4 weeks.
  Interventions: Drug: levetiracetam
- Placebo-Levetiracetam (Experimental): This group receives placebo for 4 weeks twice daily, then has a break where no treatment is given for 4 weeks, and then receives levetiracetam for 4 weeks.
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam
  Other Names: Keppra

SUMMARY:
Patients with Alzheimer's disease (AD) can have seizures in addition to losing their memory and other mental functions (referred to as cognitive functions). The seizures, and other examples of overactive electrical activity in the brain that is not noticeable, contribute to the loss of cognitive function. Studies in animal models of AD suggest that a drug that prevents seizures called levetiracetam may reduce neuronal over-excitation and improve cognition. Based on this evidence, the investigators propose to determine if levetiracetam can be used to treat patients with AD. The investigators developed novel instruments for this population that will also be used in future large-scale clinical trials.

The current study will last for 12 weeks and will involve people with AD. Participants will be initially examined with an overnight brain wave study to assess for silent epileptic (seizure-like) activity. Presence of epileptic activity on the screening exam is not required to enter the trial. Participants will then be assigned to groups in a randomized manner. One group will receive levetiracetam for 4 weeks, then no drug for 4 weeks, and then placebo for 4 weeks. For another group, the order of treatments will be reversed. The cognitive abilities of participants will be retested every 4 weeks and compared to those at the beginning. The cognitive tests include a virtual-reality navigation test of memory and computerized tests of mental flexibility and problem solving. The participants will be monitored with a magnetoencephalogram (MEG) with simultaneous EEG (M/EEG) at each visit. M/EEG is a highly effective non-invasive method for identifying brain regions of epileptic activity. The investigators will need to recruit 36 randomized participants to test the study hypotheses. This study will take place at the University of California, San Francisco (UCSF) and the University of Minnesota.

DETAILED DESCRIPTION:
For a more detailed explanation of the study and what our results were, please read our publication at https://jamanetwork.com/journals/jamaneurology/fullarticle/2784539

ELIGIBILITY:
To be included in the trial all of the following inclusion criteria must be met:

Ability to obtain written informed consent from the patient or caregiver as a surrogate; Meets National Institute on Aging-Alzheimer's Association Workgroups criteria for probable AD dementia (McKhann et al. 2011); Age ≤ 80 years at time of screening; Willing and able caregiver who has daily contact with the subject; Mini-Mental State Examination (MMSE) score ≥ 18 and/or Clinical Dementia Rating (CDR) < 2 at the initial screening assessment; Subjects and caregivers must be able to comply with prescribed regime of study treatment throughout the course of the study, and meet the required time commitment of four days of in-person visits; Any concurrent treatment for AD approved by the Food and Drug Administration (FDA), such as donepezil, galantamine, or rivastigmine, and memantine, must be stable for at least 30 days prior to screening and at least 60 days prior to study day 1. Other medications (except those listed under exclusion criteria) are allowed as long as the dose is stable for 30 days prior to screening.

The following criteria are considered grounds for exclusion:

Any conditions which could account for cognitive deficits in addition to AD, including but not limited to Vitamin B12 or folate deficiency, abnormal thyroid function, posttraumatic conditions, syphilis, multiple sclerosis or another neuroinflammatory disorder, Parkinson's disease, vascular or multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, central nervous system (CNS) tumor, progressive supranuclear palsy, subdural hematoma, etc.; Previous history of a seizure disorder, excepting cases where the first seizure or detection of epileptiform activity was within 5 years of screening and the patient is not prescribed an anticonvulsant; Significant systemic medical illnesses; Use of medications likely to affect CNS functions (e.g., benzodiazepines, narcotics); Severe renal dysfunction with creatine clearance < 30 ml/min, which would affect serum LEV levels; Participation in another AD clinical trial within 3 months of Screening, or any AD clinical trial, such as a vaccine, that has potential long-term effects; Treatment with another study drug or investigational drug within 30 days of Screening; Pregnant or lactating; Any other medical condition which is determined by the investigators to potentially create an undue risk for an adverse effect; Biomarker evidence unsupportive of a diagnosis of AD.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Vossel, MD, MSc, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - UCSF, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Background] Verret L, Mann EO, Hang GB, Barth AM, Cobos I, Ho K, Devidze N, Masliah E, Kreitzer AC, Mody I, Mucke L, Palop JJ. Inhibitory interneuron deficit links altered network activity and cognitive dysfunction in Alzheimer model. Cell. 2012 Apr 27;149(3):708-21. doi: 10.1016/j.cell.2012.02.046. PMID 22541439
- [Background] Sanchez PE, Zhu L, Verret L, Vossel KA, Orr AG, Cirrito JR, Devidze N, Ho K, Yu GQ, Palop JJ, Mucke L. Levetiracetam suppresses neuronal network dysfunction and reverses synaptic and cognitive deficits in an Alzheimer's disease model. Proc Natl Acad Sci U S A. 2012 Oct 16;109(42):E2895-903. doi: 10.1073/pnas.1121081109. Epub 2012 Aug 6. PMID 22869752
- [Background] Roberson ED, Scearce-Levie K, Palop JJ, Yan F, Cheng IH, Wu T, Gerstein H, Yu GQ, Mucke L. Reducing endogenous tau ameliorates amyloid beta-induced deficits in an Alzheimer's disease mouse model. Science. 2007 May 4;316(5825):750-4. doi: 10.1126/science.1141736. PMID 17478722
- [Background] Bakker A, Krauss GL, Albert MS, Speck CL, Jones LR, Stark CE, Yassa MA, Bassett SS, Shelton AL, Gallagher M. Reduction of hippocampal hyperactivity improves cognition in amnestic mild cognitive impairment. Neuron. 2012 May 10;74(3):467-74. doi: 10.1016/j.neuron.2012.03.023. PMID 22578498
- [Background] Vossel KA, Beagle AJ, Rabinovici GD, Shu H, Lee SE, Naasan G, Hegde M, Cornes SB, Henry ML, Nelson AB, Seeley WW, Geschwind MD, Gorno-Tempini ML, Shih T, Kirsch HE, Garcia PA, Miller BL, Mucke L. Seizures and epileptiform activity in the early stages of Alzheimer disease. JAMA Neurol. 2013 Sep 1;70(9):1158-66. doi: 10.1001/jamaneurol.2013.136. PMID 23835471
- [Background] Mares P, Mikulecka A. Different effects of two N-methyl-D-aspartate receptor antagonists on seizures, spontaneous behavior, and motor performance in immature rats. Epilepsy Behav. 2009 Jan;14(1):32-9. doi: 10.1016/j.yebeh.2008.08.013. Epub 2008 Sep 30. PMID 18786655
- [Background] Molaie M, Culebras A, Miller M. Effect of interictal epileptiform discharges on nocturnal plasma prolactin concentrations in epileptic patients with complex partial seizures. Epilepsia. 1986 Nov-Dec;27(6):724-8. doi: 10.1111/j.1528-1157.1986.tb03601.x. PMID 3780608
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Galasko D, Bennett D, Sano M, Ernesto C, Thomas R, Grundman M, Ferris S. An inventory to assess activities of daily living for clinical trials in Alzheimer's disease. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S33-9. PMID 9236950
- [Background] Schneider LS, Olin JT, Doody RS, Clark CM, Morris JC, Reisberg B, Schmitt FA, Grundman M, Thomas RG, Ferris SH. Validity and reliability of the Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S22-32. doi: 10.1097/00002093-199700112-00004. PMID 9236949
- [Background] Walker MP, Ayre GA, Cummings JL, Wesnes K, McKeith IG, O'Brien JT, Ballard CG. The Clinician Assessment of Fluctuation and the One Day Fluctuation Assessment Scale. Two methods to assess fluctuating confusion in dementia. Br J Psychiatry. 2000 Sep;177:252-6. doi: 10.1192/bjp.177.3.252. PMID 11040887
- [Background] Hinkley LB, Vinogradov S, Guggisberg AG, Fisher M, Findlay AM, Nagarajan SS. Clinical symptoms and alpha band resting-state functional connectivity imaging in patients with schizophrenia: implications for novel approaches to treatment. Biol Psychiatry. 2011 Dec 15;70(12):1134-42. doi: 10.1016/j.biopsych.2011.06.029. Epub 2011 Sep 8. PMID 21861988
- [Derived] Vossel K, Ranasinghe KG, Beagle AJ, La A, Ah Pook K, Castro M, Mizuiri D, Honma SM, Venkateswaran N, Koestler M, Zhang W, Mucke L, Howell MJ, Possin KL, Kramer JH, Boxer AL, Miller BL, Nagarajan SS, Kirsch HE. Effect of Levetiracetam on Cognition in Patients With Alzheimer Disease With and Without Epileptiform Activity: A Randomized Clinical Trial. JAMA Neurol. 2021 Nov 1;78(11):1345-1354. doi: 10.1001/jamaneurol.2021.3310. PMID 34570177
- [Derived] Liu J, Wang LN. Treatment of epilepsy for people with Alzheimer's disease. Cochrane Database Syst Rev. 2021 May 11;5(5):CD011922. doi: 10.1002/14651858.CD011922.pub4. PMID 33973646
- See also: Memory & Aging Center Website — http://memory.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on October 16,2014. Participants were recruited at the University of California, San Francisco, and the University of Minnesota, Twin Cities.
Pre-assignment Details: Participants were excluded if they were older than 80, had no diagnosis of probable AD, had a Mini-Mental State Examination score lower than 18 points or a Clinical Dementia Rating (CDR) score higher than 2 points. Patients receiving antiseizure drugs for any reason were excluded.
Groups:
- Levetiracetam-Placebo: This group receives levetiracetam for 4 weeks twice daily, then has a break where no treatment is given for 4 weeks, and then receives placebo for 4 weeks.
  levetiracetam
- Placebo-Levetiracetam: This group receives placebo for 4 weeks twice daily, then has a break where no treatment is given for 4 weeks, and then receives levetiracetam for 4 weeks.
  levetiracetam
Period: Overall Study
Arm/Group | Levetiracetam-Placebo | Placebo-Levetiracetam
Started | 17 | 17
Completed | 13 (4 Discontinued intervention because of participant's decision) | 15 (1 Discontinued intervention because of participant's decision 1 Excluded per protocol because of biomarkers inconsistent with AD)
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam-Placebo | Placebo-Levetiracetam | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 17 | 17 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Changes in Executive Function as Measured by the NIH EXAMINER Computer Battery
Description: Changes in executive function were measured using the NIH EXAMINER, a 1-hour computer-based battery of various executive function tasks. The subject's performance after the study treatment will be compared with results from a baseline assessment done before the study treatment, using statistical tests to assess whether there was any significant change. The Examiner assessment consists of the following scales: antisaccade , set shifting , flanker task, dot counting, spatial 1-back, category fluency, and letter fluency. Scores for this task have an indefinite range. Higher scores however do indicate better performance. Scores for this scale were generated using item response theory. For this study, scores with SEs greater than 0.55 were classified as unreliable and excluded from analysis. Composite scores from 2 participants were excluded on this basis.The EXAMINER ranges for the participants in the study were -2.59 to 1.33.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Levetiracetam: Those taking the test during their Levetiracetam treatment phase, whether it be before or after the crossover.
- Placebo: THose receiving placebo treatment, whether before or after the crossover.
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 22 | 22
score on a scale | -0.06 [-0.24 to 0.11] | -0.14 [-0.32 to 0.05]
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.55, ANOVA; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.18 to 0.32]

2. Secondary Outcome: Changes in Stroop Interference Naming
Description: Stroop Test - The Stroop Test (Stroop 1935) will be used to assess executive functions including selective attention, cognitive flexibility and processing speed. Subtasks include Stroop color naming and Stroop interference naming, and each subtask is restricted to 1 minute. The minimum score is 0 and the maximum score is 126. The higher the score the better a participant does.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Placebo: Those taking the test during their placebo treatment phase, whether before or after the crossover.
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 22 | 22
score on a scale | 1.5 [-1.4 to 4.3] | -1.4 [-3.6 to 0.7]
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.14, ANOVA; Mean Difference (Net) = 2.9, 95% CI 2-sided [-1.0 to 6.8]

3. Secondary Outcome: Changes in ADAS-cog
Description: Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog) - The ADAS-cog rating instrument (Rosen et al. 1984) will be used to evaluate the global cognitive functioning. The ADAS-cog is a 70-point scale that includes an assessment of verbal memory, language, orientation, reasoning, and praxis.The score is derived from adding point values from each of its subsections. The higher your score on the ADAS-cog, the better you do.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Population: 24 participants in this study did the ADAS-cog at both baseline and treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale | -0.2 [-1.8 to 1.5] | 0.8 [-0.7 to 2.3]
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = .43, ANOVA; Mean Difference (Net) = -1.0, 95% CI 2-sided [-3.4 to 1.5]

4. Secondary Outcome: Clinical Dementia Rating Sum of Boxes (CDR-SOB)
Description: Clinical Dementia Rating Sum of Boxes (CDR-SOB) - The CDR will be used as a global measure of dementia severity (Morris 1993). The CDR consists of questions addressed to the caregiver/informant. The lowest score one can receive is a 0 and the highest is a 3. Score is measured by getting the mean of the individual scores in each category. Lower scores equate to less dementia severity.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 28 | 28
score on a scale | 0.1 [-0.1 to 0.3] | 0.1 [-0.2 to 0.3]
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.63, ANOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.4]

5. Secondary Outcome: Changes in Behavior and Level of Disability - ADCS-ADL
Description: Alzheimer's Disease Cooperative Study Activities of Daily Living Scale (ADCS-ADL) - The ADCS-ADL rating instrument (Galasko et al. 1997) will be used to evaluate functional capacity. The ADCS-ADL is a caregiver rated questionnaire. Scores on the 24-item ADCS-ADL range from 0 to 78. A higher score indicates less severity while a lower score indicates greater severity.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 28 | 28
score on a scale | 0.4 [-0.9 to 1.6] | 0.3 [-0.9 to 1.5]
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.90, ANOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.1 to 1.3]

6. Secondary Outcome: Changes in Behavior and Level of Disability - ADCS-CGIC
Description: ADCS-Clinical Global Impression of Change (ADCS-CGIC) - The ADCS-CGIC is a seven-point scale that gives a global rating of change from baseline (Schneider et al. 1997). The baseline and follow up assessments are based on interviews with the subject and the informant. The ADCS-CGIC is a clinician-rated measure of: global severity at baseline scored from 1 (normal, not at all ill) to 7 (among the most extremely ill patients); and global change at follow-up scored from 1 (marked improvement) to 7 (marked worsening), where 4 indicates no change.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 28 | 28
score on a scale | 4.0 [3.8 to 4.3] | 4.0 [3.7 to 4.3]
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.80, ANOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.3 to 0.3]

7. Secondary Outcome: Changes in Behavior and Level of Disability - Neuropsychiatric Inventory (NPI)
Description: Neuropsychiatric Inventory (NPI) - The NPI (Cummings et al. 1994) will be used to evaluate the severity of behavioral symptoms. The severity scale has scores ranging from 1 to 3 points (1=mild; 2=moderate; and 3=severe) and the scale for assessing caregiver distress has scores ranging from 0 to 5 points (0=no distress; 1=minimal distress; 2=mild distress; 3=moderate distress; 4=severe distress; and 5=extreme distress).
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Levetiracetam: Those doing the interview during their Levetiracetam treatment phase, whether it be before or after the crossover.
- Placebo: Those doing the interview during their placebo treatment phase, whether before or after the crossover.
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 28 | 28
score on a scale | -0.8 [-2.7 to 1.2] | 0.2 [-2.2 to 2.6]
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.46, ANOVA; Mean Difference (Net) = -1.0, 95% CI 2-sided [-3.6 to 1.7]

8. Secondary Outcome: Changes in Epileptiform Events
Description: Epileptiform activity will be measured using a 1-hr resting magnetoencephalogram/electroencephalogram (M/EEG). M/EEG can detect abnormal epileptiform findings called "spikes". The M/EEG will be read by an epileptologist with specialized training to assess whether there are any spikes. If spikes are observed during the M/EEG they will be counted to determine their frequency (e.g., 5 spikes per 1 hour recording). The frequency of spikes will then be compared to baseline values from before beginning the study treatment, using statistical tests to determine if the frequency changed with treatment.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (95% Confidence Interval); unit: Epileptiform events
Groups:
- Levetiracetam: Activity measured during their Levetiracetam treatment phase, whether it be before or after the crossover.
- Placebo: Activity during their placebo treatment phase, whether before or after the crossover.
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 9 | 9
Epileptiform events | -0.1 [-0.4 to 0.1] | -0.2 [-1.1 to 0.6]
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.40, ANOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.9 to 1.1]

9. Other Pre Specified Outcome: Stroop Interference in AD With Epileptiform Activity
Description: Stroop Test - The Stroop Test (Stroop 1935) will be used to assess executive functions including selective attention, cognitive flexibility and processing speed. Subtasks include Stroop color naming and Stroop interference naming, and each subtask is restricted to 1 minute. The minimum score is 0 and the maximum score is 126. The higher the score the better a participant does. The mean below represents the average change in score between the timepoints for all participants.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Population: Specifically, this analysis is only looking at individuals who displayed epoileptiform activity.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Levetiracetam (Epileptiform Activity): Those with epileptiform activity taking the test during their Levetiracetam treatment phase, whether it be before or after the crossover.o.
- Placebo (Epileptiform Activity): Those with epileptiform activity taking the test during their placebo treatment phase, whether before or after the crossover.
Arm/Group | Levetiracetam (Epileptiform Activity) | Placebo (Epileptiform Activity)
Number analyzed (Participants) | 9 | 9
score on a scale | 4.7 (7.2) | -2.6 (5.0)
Statistical Analysis 1: Comparison: Levetiracetam (Epileptiform Activity) vs Placebo (Epileptiform Activity); Test type: Superiority; p = 0.046, ANOVA; Mean Difference (Net) = 7.4, 95% CI 2-sided [0.2 to 14.7]

10. Other Pre Specified Outcome: ADAS-cog in AD With Epileptiform Activity
Description: as for outcome 3
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Population: Specifically, this analysis is only looking at individuals who displayed epileptiform activity.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Levetiracetam (Epileptiform Activity): Those with epileptiform activity taking the test during their Levetiracetam treatment phase, whether it be before or after the crossover.
Arm/Group | Levetiracetam (Epileptiform Activity) | Placebo (Epileptiform Activity)
Number analyzed (Participants) | 9 | 9
score on a scale | -1.0 (4.1) | 1.5 (4.5)
Statistical Analysis 1: Comparison: Levetiracetam (Epileptiform Activity) vs Placebo (Epileptiform Activity); Test type: Superiority; p = .30, ANOVA; Mean Difference (Net) = -2.5, 95% CI 2-sided [-7.8 to 2.7]

11. Other Pre Specified Outcome: Changes in Cognitive Function as Measured by a Virtual Route Learning Test
Description: A 20-minute computer-based virtual navigation test will be used to assess how well a subject can navigate a virtual community to reach a goal destination. The subjects will then be measured on their ability to accurately navigate the virtual community after a period of a few hours. The subject's performance after the study treatment will be compared with results from a baseline assessment done before the study treatment, using statistical tests to assess whether there was any significant change.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (95% Confidence Interval); unit: correct turns
Groups:
- No Epileptiform Activity: Those who did the task without any sign of epileptiform activity.
- Epileptic Activity: Those who did the task who displayed epileptic activity
Arm/Group | No Epileptiform Activity | Epileptic Activity
Number analyzed (Participants) | 7 | 5
correct turns | -6.0 [-21.4 to 9.4] | 17.4 [-0.6 to 35.4]
Statistical Analysis 1: Comparison: No Epileptiform Activity vs Epileptic Activity; Test type: Superiority; p = 0.52, Cohen f; Mean Difference (Net) = 3.8, 95% CI 2-sided [-8.5 to 16.0]

12. Other Pre Specified Outcome: Standardized Assessments of Clinical Fluctuations -The Clinician Assessment of Fluctuation
Description: Two standardized methods will be used to quantitate fluctuations of dementia symptoms: The Clinician Assessment of Fluctuation and the One Day Fluctuation Assessment Scale (Walker et al. 2000). : The Clinician Assessment of Fluctuation (score range,0-12 points, with higher scores indicating more fluctuations),26 the One Day Fluctuation Assessment Scale (score range,0-21 points, with higher scores indicatingmore fluctuations).
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Levetiracetam: Those doing the assessment during their Levetiracetam treatment phase, whether it be before or after the crossover.
- Placebo: Those doing the activity during their placebo treatment phase, whether before or after the crossover.
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 28 | 28
score on a scale | 0.9 (2.6) | 0.1 (3.4)
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.40, ANOVA; Mean Difference (Net) = 0.7, 95% CI 2-sided [-1.0 to 2.4]

13. Other Pre Specified Outcome: Blood Serum Prolactin Level
Description: Blood samples intended for Quest Diagnostics LEV and prolactin serum levels (one 6 mL tube) will be processed in the following manner, as outlined in the Quest Diagnostics lab manual. The whole blood will be allowed to clot for 60 minutes and centrifuged at 2200 - 2500 revolutions per minute (RPM) for at least 15 minutes. The resulting serum will be split into 2 cryovials which will be stored at -20°C and immediately shipped for external assessment of LEV and prolactin levels. Prolactin will be assessed via immunoassay. The concentration of LEV in serum will be measured using validated liquid chromatography/tandem mass spectrometry (LC/MS-MS) methods.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Levetiracetam: Those who were on Leviteracetam treatment.
- Placebo: THose on placebo treatment.
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 24 | 24
ng/mL | 0.1 (1.9) | 0.2 (1.5)
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = 0.63, ANOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.1 to 0.7]

14. Other Pre Specified Outcome: NIH EXAMINER in AD With Epileptiform Activity
Description: Changes in executive function will be measured using the NIH EXAMINER, a 1-hour computer-based battery of various executive function tasks. The subject's performance after the study treatment will be compared with results from a baseline assessment done before the study treatment, using statistical tests to assess whether there was any significant change. The Examiner assessment consists of the following scales: NIH EXAMINER - antisaccade , NIH EXAMINER - set shifting , NIH EXAMINER - flanker task, NIH EXAMINER - dot counting, NIH EXAMINER - spatial 1-back, NIH EXAMINER - category fluency, and NIH EXAMINER - letter fluency. Scores for this task have an indefinite range. Higher scores however do indicate better performance. Scores for this scale were generated using item response theory (Kramer et al. J Int Neuropsychol Soc. 2014;20(1):11-19. doi:10.1017/S1355617713001094).
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Population: Specifically, this analysis is only looking at individuals who displayed epileptiform activity.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- No Epileptiform Activity: Those who took the test but displayed no evidence of epileptiform activity.
- Epileptiform Activity: THose who took the test and show evidence of epileptiform activity.
Arm/Group | No Epileptiform Activity | Epileptiform Activity
Number analyzed (Participants) | 14 | 8
score on a scale | -0.01 [-0.39 to 0.37] | 0.22 [-0.05 to 0.49]

15. Other Pre Specified Outcome: Standardized Assessments of Clinical Fluctuations - One Day Fluctuation Assessment Scale
Description: The One Day Fluctuation Assessment Scale will be used to quantitate fluctuations of dementia symptoms (Walker et al. 2000). The One Day Fluctuation Assessment Scale has a score range of 0-21 points,with higher scores indicatingmore fluctuations.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 28 | 28
score on a scale | 0.3 (1.8) | -0.4 (1.6)
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority; p = .15, ANOVA; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.3 to 1.8]

16. Other Pre Specified Outcome: MEG Power Spectrum Measures
Description: The power spectral density for different frequency bands will be measured via resting-state magnetoencephalography (MEG). A 60-second artifact-free recording segment from the first 10 minutes of recording (prior to sleep onset) will be manually selected for analysis. In participants who are able to complete additional tests, the investigators will measure dynamics of neural responses during cognitive tasks such as speech preparation and execution.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: MEG Functional Connectivity Measures
Description: Whole-brain alpha-band functional connectivity will be derived from MEG-imaging (MEG-I) using the 60-second artifact-free recording epoch that is selected for the MEG spectral analysis. MEG-I uses MEG sensor data with millisecond precision and applies source reconstruction algorithms to overlay cortical oscillatory activity onto structural brain images. Source-space MEG-I reconstructions and functional connectivity metrics will be computed with the NUTMEG software suite (http://nutmeg.berkeley.edu). The investigators will compute imaginary coherence, which is a reliable metric for functional connectivity with MEG reconstruction. Functional connectivity will measure the strength of coherence between a given region and the rest of the brain. The investigators will perform an unbiased search for MEG-I functional connectivity deficits that correlate with specific cognitive, behavioral, and functional deficits. Hinkley et al. 2011 provides details of the methodology.
Time Frame: Difference between weeks 0-4 (Baseline) and weeks 8-12 (Treatment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years, 8 months
Groups:
- Levetiracetam: Adverse events occurring when participants were taking Levetiracetam.
- Placebo: Adverse events occurring when participants were taking Placebo.
Arm/Group | Levetiracetam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 7/34 | 5/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=34) | Placebo (N=34)
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 3
Irritability (Psychiatric disorders) | 2 | 0
Tiredness (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT02002819/Prot_SAP_000.pdf